CLINICAL TRIAL: NCT01028755
Title: An Open Label Phase I Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Maximum Tolerated Dose of BAY79-4620 in Patients With Advanced Solid Tumors
Brief Title: To Determine Maximum Tolerated Dose of BAY79-4620 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12671
Record Dates: First submitted 2009-11-04; First posted 2009-12-09 (Estimated); Last update posted 2015-01-21 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasms
Keywords: Maximum Tolerated Dose
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Drug: BAY79-4620

INTERVENTIONS:
Drug: BAY79-4620 — BAY79-4620 will be administered as 1 hour IV infusion. Dose escalation will be dependent on any dose limiting toxicities

SUMMARY:
This is the first time this drug will be tested in humans in order to determine the safety of the drug, the ability to tolerate the drug, to measure how the drug is used in the body and as a result of these tests to determine a maximum dose to be given. Specifically, the following aspects will be investigated:

* side effects of BAY79-4620 given as infusion every three weeks
* evaluation of highest and safest dose of BAY79-4620
* distribution and concentration of BAY79-4620 in the blood at specific times after administration
* effect of BAY79-4620 on tumor growth
* assessment of "biomarkers" (eg, analysis of specific proteins in blood samples, or analysis of tumor tissue sampled at the time of cancer diagnosis) for changes during the treatment or prediction of safety or benefits of the treatment with BAY79-4620.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than/equal to 18 years old.
* ECOG Performance Status of 0 - 2
* Life expectancy of at least 12 weeks
* Patients with advanced, histologically or cytological confirmed solid tumors, refractory to any standard therapy or have no standard therapy available
* Radiographically or clinically evaluable tumor
* Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements to be conducted within 14 days prior to start of first dose:
* Hemoglobin > 10.0 g/dL
* Absolute neutrophil count (ANC) > or = 1500/mm3
* Platelet count > or = 100,000 /mm3
* Total bilirubin < or = 1.5 times the upper limit of normal
* ALT and AST < or = 2.5 x upper limit of normal (< or = 5 x upper limit of normal for patients with liver involvement)
* INR less than or = 1.5 and a PTT within normal limits (patients who do not undergo an anticoagulative treatment, but have an abnormal high PTT while INR is normal, indicating towards an artificial PTT elevation caused by heparinized, are eligible.
* Serum creatinine < 1.5 times the upper limit of normal

Exclusion Criteria:

* History of impaired cardiac function or clinically significant cardiac disease (i.e. congestive heart failure (CHF) NYHA Class III or IV); myocardial infarction, unstable angina or cardiac arrhythmias requiring anti-arrhythmic therapy < 6 months prior to study entry (beta blockers or digoxin are permitted) and LVEF <40% (as measured at screening by MUGA or echocardiogram).
* Patients with amylase or lipase greater than upper limit of normal range per local laboratory
* History of pancreatitis
* Uncontrolled hypertension defined as systolic blood pressure > 150 mm Hg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management
* Symptomatic metastatic brain or meningeal tumors unless the patient is > 6 months from definitive therapy, has no evidence of tumor growth on an imaging study within 2 weeks prior to study entry, and is clinically stable with respect to the tumor at the time of study entry.
* Patients with severe renal impairment or on dialysis
* Known human immunodeficiency virus (HIV) infection or patients with an active hepatitis B or C infection necessitating treatment. Patients with chronic hepatitis B or C are eligible
* Active clinically serious infections > CTCAE Grade 2
* Serious, non-healing wound, ulcer, or bone fracture
* Known or suspected allergy or intolerance to any agent given in the course of this trial
* Previous cancer that is distinct in primary site or histology from actual disease EXCEPT cervical cancer in-situ, treated basal cell carcinoma, superficial bladder tumors [Ta and Tis] or any cancer curatively treated > 3 years prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-11; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability, maximum tolerated dose | 2 years
Pharmacokinetics profile of BAY79-4620 and its key metabolites | 2 years

SECONDARY OUTCOMES:
Biomarker evaluation | 2 years
Tumor response | 2 years
Immunogenicity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (2):
- United States (2):
  - Nashville, Tennessee
  - San Antonio, Texas